CLINICAL TRIAL: NCT04141462
Title: EXOME Analysis Position in the Strategy of Genetic Predisposition Factors Identification in Early-onset Cancer
Acronym: EX²TRICAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EX²TRICAN
Record Dates: First submitted 2019-10-23; First posted 2019-10-28 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Cancer; Genetic Predisposition
Keywords: genetic mutations; early sporadic or familial cancer; gene panel; exome analysis; high-throughput exome sequencing
MeSH Terms: conditions — Neoplasms; Genetic Predisposition to Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with a a constitutional genetic alteration (Experimental): one genetic consultation and one blood test
  Interventions: Genetic: blood sample

INTERVENTIONS:
Genetic: blood sample — blood test

SUMMARY:
5 to 10% of cancers are due to the presence of a constitutional genetic alteration. It can be inherited from parents (family form) or by accident, in the first moments of life after fertilization (sporadic form). In both cases, this genetic alteration is constitutional and transmissible to descendants. It is hereditary. When an hereditary early form is suspected, several well-known genes generally involved in genetic predispositions to cancer are found by a technique called " gene panel ". However, this analysis does not always identify the genetic predisposing factors for cancer. New techniques called "high-throughput exome sequencing (SHD-E)", allow more than the analysis of the the gene panel. These analysis allow to identify alterations in other genes that could contribute to the development of cancer. The objective of the Ex²trican study is to show, from patients with early cancer (sporadic or familial form), that this approach to exome sequencing can be effective to identify new genetic risk of cancer, when the first panel analysis of genes is negative.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the interest of the SHD-E approaches after a negative result of the analysis called " gene panel " tested in routine in order to identify a genetic factor of predisposition to the cancer.

ELIGIBILITY:
Inclusion Criteria:

Index case:

1. Major or minor patient
2. Histological or cytological evidence of malignant tumor diagnosis
3. Patient with cancer before age 40 (or before age 30 for breast cancer).
4. Absence of anomaly found on the oncogenetic panel tested in the predisposition concerned
5. Patient affiliated to a social security scheme
6. Signature of Informed Consent EXTRICAN
7. Availability of a tumor sample if needed secondary functional studies
8. Availability of both parents when the trio approach will be necessary in the population 1 (or validation of the indication in CPR in case of non-availability of both parents)
9. Availability of affected relatives in population 2 (or validation of the indication in SPC in case of non-availability of the related person)

Related:

1. Major or minor patient
2. Histological or cytological evidence of the diagnosis of malignant tumor if
3. Patient affiliated to a social security scheme
4. Signing informed consent EXTRICAN

Exclusion Criteria:

Index and related case:

1. Refusal of the patient participation
2. Psychiatric illness and / or condition of the patient compromising the understanding of the information or the realization of the study
3. Patient under guardianship, curatorship or safeguard of justice
4. Pregnant woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2026-04-07 (Estimated); Study Completion 2028-04-07 (Estimated)

PRIMARY OUTCOMES:
genetic mutations | inclusion
  SHD-E analysis

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHRU Jean Minjoz, Besançon
  - Centre Georges-François Leclerc, Dijon
  - CHU de Dijon, Dijon
  - CHU de Reims, Reims
  - Polyclinique de Courlancy, Reims
  - CH de Troyes, Troyes